CLINICAL TRIAL: NCT05761860
Title: The Potential of Oxytocin to Reduce Opioid Abuse Liability and Pain Among Older Adults
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202300435; 5R21DA056813-02 (NIH)
Record Dates: First submitted 2023-02-27; First posted 2023-03-09 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Pain
Keywords: Pain; Abuse liability
MeSH Terms: conditions — Pain | interventions — Oxycodone; Tablets

STUDY DESIGN:
Intervention Model Description: This is a within-participant study so that each participant receives all conditions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Oral oxycodone (5mg) + intranasal oxytocin (48 IU) (Active Comparator): Combined effects of oxycodone and oxytocin.
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Drug: Oxytocin Nasal Spray (48 IU)
- Oral oxycodone (2.5mg) + intranasal oxytocin (48 IU) (Active Comparator): Combined effects of oxycodone and oxytocin.
  Interventions: Drug: OxyCODONE 2.5 mg Oral Tablet; Drug: Oxytocin Nasal Spray (48 IU)
- Oral placebo + intranasal oxytocin (48 IU) (Active Comparator): Separate effects of oxytocin. As is standard methodology in abuse liability and pain assessments, a placebo condition will be included for each drug in order to compare the abuse liability and pain assessments change from placebo.
  Interventions: Other: Placebo oxyCODONE Oral Tablet; Drug: Oxytocin Nasal Spray (48 IU)
- Oral oxycodone (5mg) + intranasal placebo (Active Comparator): Separate effects of oxycodone. As is standard methodology in abuse liability and pain assessments, a placebo condition will be included for each drug in order to compare the abuse liability and pain assessments change from placebo.
  Interventions: Drug: OxyCODONE 5 mg Oral Tablet; Other: Placebo Oxytocin Nasal Spray
- Oral oxycodone (2.5mg) + intranasal placebo (Active Comparator): Separate effects of oxycodone. As is standard methodology in abuse liability and pain assessments, a placebo condition will be included for each drug in order to compare the abuse liability and pain assessments change from placebo.
  Interventions: Drug: OxyCODONE 2.5 mg Oral Tablet; Other: Placebo Oxytocin Nasal Spray
- Oral placebo + intranasal placebo (Sham Comparator): Serves as the control.
  Interventions: Other: Placebo oxyCODONE Oral Tablet; Other: Placebo Oxytocin Nasal Spray

INTERVENTIONS:
Drug: OxyCODONE 5 mg Oral Tablet — Oxycodone 5mg oral administration
  Arms: Oral oxycodone (5mg) + intranasal oxytocin (48 IU); Oral oxycodone (5mg) + intranasal placebo
Drug: OxyCODONE 2.5 mg Oral Tablet — Oxycodone 2.5mg oral administration
  Arms: Oral oxycodone (2.5mg) + intranasal oxytocin (48 IU); Oral oxycodone (2.5mg) + intranasal placebo
Other: Placebo oxyCODONE Oral Tablet — Oxycodone 0mg (placebo) oral administration
  Arms: Oral placebo + intranasal oxytocin (48 IU); Oral placebo + intranasal placebo
Drug: Oxytocin Nasal Spray (48 IU) — Intranasal oxytocin administration (48 IU)
  Arms: Oral oxycodone (2.5mg) + intranasal oxytocin (48 IU); Oral oxycodone (5mg) + intranasal oxytocin (48 IU); Oral placebo + intranasal oxytocin (48 IU)
Other: Placebo Oxytocin Nasal Spray — Intranasal oxytocin placebo administration
  Arms: Oral oxycodone (2.5mg) + intranasal placebo; Oral oxycodone (5mg) + intranasal placebo; Oral placebo + intranasal placebo

SUMMARY:
Some research suggests that administration of oxytocin with oxycodone may reduce its abuse liability and improve its ability to reduce pain. In a 6-session laboratory study, we will be evaluating the effects of oxycodone and oxytocin (combined and separately, across sessions) on experimentally-induced pain, subjective effects, and decision-making.

DETAILED DESCRIPTION:
The overall project goals are to determine oxytocin effects on oxycodone's subject-rated abuse liability, and experimental pain. Generally healthy individuals (determined via medical history review and a screening session) will, after informed consent, self-administer intranasal oxytocin (or placebo, containing the same ingredients but no oxytocin) shortly after oral oxycodone or placebo in a non-residential, double-blind, randomized, placebo-controlled, within-subjects laboratory study. Prescreening will assure drug application safety and, using a validated, comprehensive pain history interview, determine previous or existing chronic pain conditions, including current pain medication use.

ELIGIBILITY:
Inclusion Criteria:

* Individuals fluent in English will participate.
* Must report some experience with opioids (e.g., oxycodone, defined as use at least once in the subject's lifetime).
* Be within 20% of their ideal body weight.
* Are not currently experiencing chronic pain (pain on most days during the past 3 months)
* Have a systolic blood pressure of <=140 and diastolic blood pressure of <= 90, and a heart rate <= 90 beats per minute.
* Participants must also have a normal electrocardiogram (EKG) reading and bloodwork indicating no major health contraindications.

Exclusion Criteria:

* Significant current physical disease or major (uncontrolled) psychiatric disorder.
* No self-reported current interest in drug abuse treatment.
* Women who are pregnant or nursing.
* Any severe comorbid illicit substance use disorders or current clinically significant withdrawal for any abused drug excluding nicotine and caffeine.

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Subject-rated abuse liability | Up to 6 weeks
  Using a Visual Analog Scale with scoring as 0=not at all, 20=possibly mild, 40=definitely mild, 60=moderately, 80=strongly, and 100=extremely, or any number in between. Testing occurs only in the context of 6 sessions due to a minimum of a one week washout period in between each session.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith S Berry, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No